CLINICAL TRIAL: NCT01697345
Title: Breast Cancer, Aromatase Inhibitor Therapy, and Sexual Functioning: A Pilot Study on the Effects of Vaginal Testosterone Therapy
Brief Title: Breast Cancer, Aromatase Inhibitor Therapy, and Sexual Functioning: The Effects of Vaginal Testosterone Therapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Melissa Dahir, Principal Investigator, Creighton University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MelissaDahir
Record Dates: First submitted 2012-09-26; First posted 2012-10-02 (Estimated); Results first posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer; Vaginal Dryness; Dyspareunia; Sexual Health Quality of Life
Keywords: Vaginal Testosterone; Vaginal atrophy; Female Sexual Dysfunction; Aromatase Inhibitors
MeSH Terms: conditions — Breast Neoplasms; Dyspareunia | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal Testosterone (Experimental): Testosterone USP micronized powder supplied by Medisca Pharmacy will be compounded by Precision Compounding pharmacy as testosterone 0.3% per 0.5 milliliters (mL) in pharmabase cream. The compounded testosterone vaginal cream will be supplied in pre-filled syringes and each 0.5 mL dose will deliver 300 mcg of testosterone daily. The cream will be applied to the vaginal opening once daily for four weeks (28 days).
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone

SUMMARY:
It is well documented that women who have breast cancer may experience a decrease in quality of life and sexual functioning due to side effects from adjuvant endocrine therapy, typically aromatase inhibitors (AIs). Women taking AIs are more likely to report unpleasant urogenital and vaginal symptoms due to the physiologic suppression of estradiol. This treatment can impair sexual functioning and cause a decreased sexual health quality of life.

At the present time, there are no Food and Drug Administration (FDA) approved medications for the vulvovaginal or sexual side effects related to the use of AIs. The lack of treatment options is concerning because the number of women diagnosed with breast cancer continues to increase; their longevity, also, continues to increase with the use of newer adjuvant chemotherapies. Local health care practitioners have observed that the benefits of vaginal testosterone for sexual health in breast cancer survivors are similar to the benefits of vaginal estrogen in women without breast cancer.

The purpose of this study is to evaluate the impact of using a daily compounded vaginal testosterone cream for 4 weeks (28 days) on breast cancer survivor's reported experience of vulvovaginal symptoms accompanying the use of AIs and their associated quality of life and sexual functioning.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer
* Currently taking an aromatase inhibitor (AI)
* Age > 50 years of age
* Postmenopausal, or two years since last menstrual cycle
* Urogenital/vulvovaginal symptoms such as vaginal dryness and pain with intercourse
* Changes in sexual health quality of life/sexual functioning since starting AI therapy

Exclusion Criteria:

* The use of other treatments for breast cancer such as chemotherapy or radiation within the past 12 months
* A known sensitivity to medications containing testosterone
* The use of exogenous hormone replacement therapy (HRT) in the past three months, including systemic and local estrogen or testosterone therapy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Dahir, DNP, Principal Investigator — Creighton University; Dianne Travers-Gustafson, PhD, Study Chair — Creighton University; Robert Langdon, MD, Study Director — Nebraska Cancer Specialists
Locations (1):
- Nebraska Cancer Specialists/Midwest Cancer Center - Legacy, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were prospectively recruited from Nebraska Cancer Specialists in Omaha, NE, between January 11, 2013, and April 23, 2013.
Pre-assignment Details: During the first study visit, the the PI procured a vaginal swab because women with suppressed estrogen levels have an increased risk for infection. Also, in the clinical setting, the PI has observed that women who develop a yeast or bacterial infection while using vaginal testosterone frequently report symptoms of vaginal burning or irritation.
Period: Overall Study
Arm/Group | Vaginal Testosterone
Started | 13
Completed | 12 (One patient withdrew due to symptoms of recurrent Gardnerella vaginalis.)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: One patient withdrew due to symptoms of recurrent Gardnerella vaginalis.
Arm/Group | Vaginal Testosterone
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.67 (6.095)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Marital Status [Number; unit: Participants]
  Married | 12
  Not Married | 0
Length of Marriage [Number; unit: participants]
  0-5 years | 1
  6-10 years | 0
  11-15 years | 0
  16-20 years | 0
  21-25 years | 5
  26-30 years | 1
  31-35 years | 2
  36-40 years | 2
  41-50 years | 0
  51-55 years | 1
Highest Level of Education [Number; unit: Participants]
  High school degree | 3
  Associate's degree | 3
  Bachelor's degree | 4
  Master's degree | 2
Oophorectomy [Number; unit: Participants]
  Yes | 4
  No | 8
Estrogen-receptor (ER) Status [Number; unit: Participants]
  ER+ | 11
  ER- | 1
Progesterone-receptor (PR) Status [Number; unit: Participants]
  PR+ | 10
  PR- | 2
Human Epidermal Growth Factor Receptor 2 (HER2) Status [Number; unit: Participants]
  HER2+ | 1
  HER2- | 11
Aromatase Inhibitor [Number; unit: Participants]
  anastrozole (Arimidex) | 11
  letrozole (Femara) | 1
  exemestane (Aromasin) | 0
Vaginal Swab Test [Number; unit: Participants] — A vaginal swab was obtained prior to prescribing testosterone therapy because women with suppressed estrogen levels have an increased risk of infection.
  Participants
    No vaginal infection | 9
    Gardnerella vaginalis | 3
    Candidiasis species | 0
Sexually Active Prior to Study [Number; unit: Participants]
  Yes | 7
  No | 5
Sexually Active During Study [Number; unit: Participants]
  Yes | 11
  No | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Female Sexual Function Index (FSFI) Score
Description: The Female Sexual Function Index (FSFI) questionnaire was administered to participants prior to starting vaginal testosterone therapy and the survey was repeated after using the study drug for 4 weeks. The participants served as their own controls. The FSFI assesses six domains of sexual functioning (desire, arousal, lubrication, orgasm, satisfaction, and pain) over the past 4 weeks. The sum of all domain scores equals the total FSFI score. The total FSFI score ranges from 2-36 and a total FSFI score < 26.5 suggests female sexual dysfunction.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FSFI Total Score (Pretest): Administered to participants prior to starting vaginal testosterone therapy.
- FSFI Total Score (Postteset): Testosterone USP micronized powder supplied by Medisca Pharmacy was compounded by Precision Compounding pharmacy as testosterone 0.3% per 0.5 milliliters (mL) in pharmabase cream. The compounded testosterone vaginal cream was supplied in pre-filled syringes and each 0.5 mL dose delivered 300 mcg of testosterone daily. The cream was applied to the vaginal opening once daily for four weeks (28 days).
Arm/Group | FSFI Total Score (Pretest) | FSFI Total Score (Postteset)
Number analyzed (Participants) | 12 | 12
units on a scale | 8.691 (3.803) | 18.783 (7.050)
Statistical Analysis 1: Comparison: FSFI Total Score (Pretest) vs FSFI Total Score (Postteset); Test type: Superiority or Other; p < 0.0005, t-test, 2 sided; Mean Difference (Final Values) = -10.092, 95% CI 2-sided [-13.928 to -6.256], Standard Deviation 6.0378

2. Primary Outcome: FSFI Desire Domain
Description: The desire score is calculated by adding the individual scores from the desire domain (question #1 and #2) and multiplying the sum by the domain factor of 0.6. The domain score for desire ranges from 1.2 (minimum) to 6 (maximum) and a higher value represents a better outcome.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FSFI Desire Domain Score (Pretest): Administered to participants prior to starting vaginal testosterone therapy.
- FSFI Desire Domain Score (Posttest): Testosterone USP micronized powder supplied by Medisca Pharmacy was compounded by Precision Compounding pharmacy as testosterone 0.3% per 0.5 milliliters (mL) in pharmabase cream. The compounded testosterone vaginal cream was supplied in pre-filled syringes and each 0.5 mL dose delivered 300 mcg of testosterone daily. The cream was applied to the vaginal opening once daily for four weeks (28 days).
Arm/Group | FSFI Desire Domain Score (Pretest) | FSFI Desire Domain Score (Posttest)
Number analyzed (Participants) | 12 | 12
units on a scale | 1.350 (0.373) | 2.650 (0.866)
Statistical Analysis 1: Comparison: FSFI Desire Domain Score (Pretest) vs FSFI Desire Domain Score (Posttest); Test type: Superiority or Other; p < 0.0005, t-test, 2 sided; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-1.859 to -0.741], Standard Deviation 0.880

3. Primary Outcome: FSFI Arousal Domain
Description: The arousal score is calculated by adding the individual scores from the arousal domain (question #3, #4, #5, #6) and multiplying the sum by the domain factor of 0.3. The arousal domain score ranges from 0 (minimum) to 6 (maximum)and a higher value represents a better outcome.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FSFI Arousal Domain Score (Pretest): Administered to participants prior to starting vaginal testosterone therapy.
- FSFI Arousal Domain Score (Posttest): Testosterone USP micronized powder supplied by Medisca Pharmacy was compounded by Precision Compounding pharmacy as testosterone 0.3% per 0.5 milliliters (mL) in pharmabase cream. The compounded testosterone vaginal cream was supplied in pre-filled syringes and each 0.5 mL dose delivered 300 mcg of testosterone daily. The cream was applied to the vaginal opening once daily for four weeks (28 days).
Arm/Group | FSFI Arousal Domain Score (Pretest) | FSFI Arousal Domain Score (Posttest)
Number analyzed (Participants) | 12 | 12
units on a scale | 1.200 (0.677) | 2.825 (1.256)
Statistical Analysis 1: Comparison: FSFI Arousal Domain Score (Pretest) vs FSFI Arousal Domain Score (Posttest); Test type: Superiority or Other; p = 0.002, t-test, 2 sided; Median Difference (Final Values) = -1.625, 95% CI 2-sided [-2.495 to -0.755], Standard Deviation 1.369

4. Primary Outcome: FSFI Lubrication Domain
Description: The lubrication score is calculated by adding the individual scores from the lubrication domain (question #7, #8, #9, #10) and multiplying the sum by the domain factor of 0.3. The domain score for lubrication ranges from 0 (minimum) to 6 (maximum) and a higher value represents a better outcome.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FSFI Lubrication Domain Score (Pretest): Administered to participants prior to starting vaginal testosterone therapy.
- FSFI Lubrication Domain Score (Posttest): Testosterone USP micronized powder supplied by Medisca Pharmacy was compounded by Precision Compounding pharmacy as testosterone 0.3% per 0.5 milliliters (mL) in pharmabase cream. The compounded testosterone vaginal cream was supplied in pre-filled syringes and each 0.5 mL dose delivered 300 mcg of testosterone daily. The cream was applied to the vaginal opening once daily for four weeks (28 days).
Arm/Group | FSFI Lubrication Domain Score (Pretest) | FSFI Lubrication Domain Score (Posttest)
Number analyzed (Participants) | 12 | 12
units on a scale | 1.175 (0.620) | 2.675 (1.929)
Statistical Analysis 1: Comparison: FSFI Lubrication Domain Score (Pretest) vs FSFI Lubrication Domain Score (Posttest); Test type: Superiority or Other; p = 0.018, t-test, 2 sided; Mean Difference (Final Values) = -1.500, 95% CI 2-sided [-2.692 to -0.308], Standard Deviation 1.876

5. Primary Outcome: FSFI Orgasm Domain
Description: The orgasm score is calculated by adding the individual scores from the orgasm domain (question #11, #12, #13) and multiplying the sum by the domain factor of 0.4. The domain score for orgasm ranges from 0 (minimum) to 6 (maximum) and a higher value represents a better outcome.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FSFI Orgasm Domain Score (Pretest): Administered to participants prior to starting vaginal testosterone therapy.
- FSFI Orgasm Domain Score (Posttest): Testosterone USP micronized powder supplied by Medisca Pharmacy was compounded by Precision Compounding pharmacy as testosterone 0.3% per 0.5 milliliters (mL) in pharmabase cream. The compounded testosterone vaginal cream was supplied in pre-filled syringes and each 0.5 mL dose delivered 300 mcg of testosterone daily. The cream was applied to the vaginal opening once daily for four weeks (28 days).
Arm/Group | FSFI Orgasm Domain Score (Pretest) | FSFI Orgasm Domain Score (Posttest)
Number analyzed (Participants) | 12 | 12
units on a scale | 1.733 (1.767) | 2.933 (2.049)
Statistical Analysis 1: Comparison: FSFI Orgasm Domain Score (Pretest) vs FSFI Orgasm Domain Score (Posttest); Test type: Superiority or Other; p = 0.005, t-test, 2 sided; Mean Difference (Final Values) = -1.20000, 95% CI 2-sided [-1.95080 to -.44920], Standard Deviation 1.18168

6. Primary Outcome: FSFI Satisfaction Domain
Description: The satisfaction score is calculated by adding the individual scores from the satisfaction domain (question #14, #15, #16) and multiplying the sum by the domain factor of 0.4. The satisfaction domain score ranges from 0.8 (minimum) to 6 (maximum) and a higher value represents a better outcome.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FSFI Satisfaction Domain Score (Pretest): Administered to participants prior to starting vaginal testosterone therapy.
- FSFI Satisfaction Domain Score (Posttest): Testosterone USP micronized powder supplied by Medisca Pharmacy was compounded by Precision Compounding pharmacy as testosterone 0.3% per 0.5 milliliters (mL) in pharmabase cream. The compounded testosterone vaginal cream was supplied in pre-filled syringes and each 0.5 mL dose delivered 300 mcg of testosterone daily. The cream was applied to the vaginal opening once daily for four weeks (28 days).
Arm/Group | FSFI Satisfaction Domain Score (Pretest) | FSFI Satisfaction Domain Score (Posttest)
Number analyzed (Participants) | 12 | 12
units on a scale | 2.300 (1.311) | 4.200 (1.293)
Statistical Analysis 1: Comparison: FSFI Satisfaction Domain Score (Pretest) vs FSFI Satisfaction Domain Score (Posttest); Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.900, 95% CI 2-sided [-2.761 to -1.039], Standard Deviation 1.355

7. Primary Outcome: FSFI Pain Domain
Description: The score for pain is calculated by adding the individual scores from the pain domain (question #17, #18, #19) and multiplying the sum by the domain factor of 0.4. The domain score for pain ranges from 0 (minimum) to 6 (maximum) and a higher value represents a better outcome.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FSFI Pain Domain Score (Pretest): Administered to participants prior to starting vaginal testosterone therapy.
- FSFI Pain Domain Score (Posttest): Testosterone USP micronized powder supplied by Medisca Pharmacy was compounded by Precision Compounding pharmacy as testosterone 0.3% per 0.5 milliliters (mL) in pharmabase cream. The compounded testosterone vaginal cream was supplied in pre-filled syringes and each 0.5 mL dose delivered 300 mcg of testosterone daily. The cream was applied to the vaginal opening once daily for four weeks (28 days).
Arm/Group | FSFI Pain Domain Score (Pretest) | FSFI Pain Domain Score (Posttest)
Number analyzed (Participants) | 12 | 12
units on a scale | 0.933 (0.875) | 3.500 (2.276)
Statistical Analysis 1: Comparison: FSFI Pain Domain Score (Pretest) vs FSFI Pain Domain Score (Posttest); Test type: Superiority or Other; p < 0.0005, t-test, 2 sided; Mean Difference (Final Values) = -2.567, 95% CI 2-sided [-3.706 to -1.428], Standard Deviation 1.793

8. Secondary Outcome: Number of Participants Who Continued Vaginal Testosterone Upon Completion of the Study
Time Frame: After 4 weeks
Measure: Number; unit: participants
Groups:
- Continued Vaginal Testosterone Therapy: Participants who chose to continue vaginal testosterone therapy upon completion of the study.
- Did Not Continue Vaginal Testosterone Therapy: Participants who chose not to continue vaginal testosterone upon completion of the study.
Arm/Group | Continued Vaginal Testosterone Therapy | Did Not Continue Vaginal Testosterone Therapy
Number analyzed (Participants) | 12 | 12
participants | 11 | 1

ADVERSE EVENTS:
Arm/Group | Vaginal Testosterone
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

LIMITATIONS AND CAVEATS:
Limitations of this pilot study included the narrow time frame for enrollment, the exclusion of surgically menopausal women under the age of 50, and symptoms of recurrent Gardnerella vaginalis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No